CLINICAL TRIAL: NCT06136247
Title: Integrating Brain, Neurocognitive, and Computational Tools in Opioid Use Disorder (OUD) to Characterize Executive Function and to Predict Clinical Outcomes.
Brief Title: Integrating Brain, Neurocognitive, and Computational Tools in OUD
Status: Recruiting | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Other Study IDs: 854332
Record Dates: First submitted 2023-11-01; First posted 2023-11-18 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Opioid Use Disorder
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Healthy controls: Healthy controls, people not living with opioid use disorder or on medication assisted therapy for such.
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: fNIRS
- Patients living with Opioid Use Disorder: Individuals with opioid use disorder who have been on a stable dose of medication assisted therapy for at least a week.
  Interventions: Diagnostic Test: Neurocognitive battery; Diagnostic Test: fNIRS

INTERVENTIONS:
Diagnostic Test: Neurocognitive battery — The Penn Computerized Neurobehavioral Battery (CNB) consists of a series of cognitive tasks, measuring accuracy and speed of performance in major cognitive domains, including executive functions (i.e., abstraction, sustained attention, working memory), episodic memory (i.e., verbal, facial, and spatial memory), complex cognitive processing (i.e., language reasoning, nonverbal reasoning, spatial processing), social cognition (i.e., emotion identification, emotion intensity differentiation, age differentiation) and processing speed (i.e., sensorimotor and motor).
Diagnostic Test: fNIRS — Functional near-infrared spectroscopy (fNIRS) is a noninvasive optical imaging technique that measures changes in oxygenated and deoxygenated hemoglobin (Hb) concentrations within the brain by means of their characteristic absorption spectra of the wavelengths range of 700-1000 nm [35,36].

SUMMARY:
The 5-year K01 Mentored Research Scientist proposal will employ brain, neurocognitive, and computational tools (e.g., machine learning) to understand the impact of opioid-use disorder (OUD) and common co-occurring issues on executive function and clinical outcomes. There have been record numbers of fatal and non-fatal overdoses (ODs) associated with opioids (and other drugs) in the past 12-months. Improving classification and predictive capabilities to enhance treatment and prevent relapse is of the upmost importance. Deficits in neurocognition often are associated with poor treatment outcomes (e.g., more drug use, medication non-adherence), yet co-occurring issues associated with OUD (e.g., depression, anxiety, physical/sexual abuse, neglect) make it difficult to parse which contributing factors lead to worse executive function (EF) and poorer treatment outcomes. Novel brain, neurocognitive, and computational tools are needed to help determine these differences, in order to lay the foundation for better treatments. This need has shaped both the training plan and the associated research project in a 5-year K01 Mentored Research Scientist proposal, building on Dr. Regier's prior preclinical and clinical addiction neuroscience experience (focused mostly on cocaine-use disorders, cue-reactivity, subcortical networks, prior adversity, and univariate imaging techniques).

ELIGIBILITY:
Inclusion Criteria:

* men and women with moderate to severe opioid use disorder by Diagnostic and Statistical Manual, version 5, (DSM-V) criteria on a stable (at least one week without change) dose of oral buprenorphine-naloxone or methadone. (for OUD group)
* Eligible participants will be between 18-60 years of age;
* able to read at an eighth-grade level;
* able to speak English.

Exclusion Criteria:

* unable to understand or complete the tasks.
* Certain mental health conditions, including (but not limited to) bipolar I with current manic episode, schizophrenia, and schizoaffective disorder, determined by the Principal Investigator (PI) to interfere with study participation.
* moderate or severe substance-use disorder (for Healthy Controls)

Ages: 18 Years to 60 Years | Sex: All
Age Groups: Adult
Study Population: 96 individuals living with OUD and on stable MAT, as well as 96 individuals who are considered healthy controls, all living in the greater Philadelphia area and able to attend study visits at the University of Pennsylvania.
Sampling Method: Non-Probability Sample
Enrollment: 192 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-07-31 (Estimated)

PRIMARY OUTCOMES:
Drug use | weeks 1 through 8
  Patient self report of drug use on the weekly Follow Up Survey- days per week having taken any drugs
Medication adherence | weeks 1 through 8
  Patient self report of medication-assisted treatment (MAT) adherence on the weekly Follow Up Survey - days per week having taken their MAT
Mental health symptoms | weeks 1 through 8
  Patient self report of mental health symptoms on the weekly Follow Up Survey - days per week of experiencing symptoms of depression or anxiety

CONTACTS AND LOCATIONS:
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No